CLINICAL TRIAL: NCT00123266
Title: An Open-label, Clinical Trial of Intra-arterial Microplasmin Administration in Patients With Acute Intracranial Vertebrobasilar Artery Occlusion
Brief Title: Intra-arterial Microplasmin Administration in Patients With Acute Intracranial Vertebrobasilar Artery Occlusion
Acronym: MITI-IA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision not to pursue development of uPLi for vascular conditions.
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG-M-003
Record Dates: First submitted 2005-07-21; First posted 2005-07-22 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Stroke
Keywords: stroke; vertebrobasilar; basilar; Acute vertebrobasilar artery occlusion
MeSH Terms: conditions — Stroke | interventions — microplasmin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active (Experimental)
  Interventions: Drug: Microplasmin

INTERVENTIONS:
Drug: Microplasmin — 2 mg/kg, IA over 75 mins

SUMMARY:
The purpose of the trial is to evaluate the safety of microplasmin as well as its ability to open blocked arteries to the brain in patients with acute stroke when given into the artery at the site of the blockage.

DETAILED DESCRIPTION:
Patients with angiographically documented acute intracranial vertebrobasilar artery occlusion presenting within 24 hours of neurological symptom onset will be enrolled into this open-label trial. During study drug administration, angiograms will be repeated at regular intervals to determine degree of clot lysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with angiographically documented vertebrobasilar artery occlusion
2. Initiation of study drug treatment within 24 hours of the onset of neurological symptoms
3. Age 18-75 (inclusive).

Exclusion Criteria:

1. Patients with coma > 6 hrs duration and complete loss of brain stem reflexes (corneal reflex, gag reflex, VOR, pupil reflexes) as measured at the last assessment before sedation/intubation
2. Rapidly improving neurologic signs at any time before initiation of study drug administration.
3. Known contrast agent-sensitivity
4. Uncontrolled hypertension defined as a systolic blood pressure > 180 mm Hg or a diastolic blood pressure > 100 mm Hg on 3 separate occasions at least 10 minutes apart or requiring continuous IV therapy.
5. History of stroke within the previous 6 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-12; Primary Completion 2007-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Recanalization rate | Day-7, Day-30 and Day-90

SECONDARY OUTCOMES:
Clinical assessment | Day-7, Day-30 and Day-90

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hamann, Prof. Dr, Principal Investigator — HSK Dr. Horst Schmidt Hospital
Locations (7):
- Germany (6):
  - UniversitÃ¤tsklinikum Erlangen, Erlangen
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - UniversitÃ¤tsklinikum des Saarlandes, Homburg/Saar
  - UKSH Campus Kiel, Kiel
  - Ludwig-Maximilians-University Hospital, Munich
  - HSK Dr. Horst Schmidt Hospital, Wiesbaden
- Sint Antonius Ziekenhuis, Nieuwegein, Netherlands